CLINICAL TRIAL: NCT03387046
Title: Evaluation of clINical reCovery After a Relapse: a Pilot Study assEssing the Neuronal Effects of D-Aspartate in RR-MS Subjects Treated With IntErferon Beta 1a 44 mcg TIW (INCREASE)
Brief Title: A Pilot Study in Participants With Relapsing Remitting Multiple Sclerosis (RR-MS)
Acronym: INCREASE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was terminated early due to slow recruitment rate.
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MS200136_0041
Record Dates: First submitted 2017-12-22; First posted 2017-12-29 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Relapsing remitting multiple sclerosis; D-Aspartate; interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — D-Aspartic Acid; peginterferon beta-1a; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-aspartate + IFN beta-1a + Methylprednisolone (Experimental): Participants received D-aspartate 2660 milligrams (mg) once daily in the form of oral solution for 24 weeks along with IFN beta-1a subcutaneously (sc) at a dose of 44 microgram (mcg) three times a week (TIW) in participants without relapse and IFN beta-1a sc TIW plus Methylprednisolone 1000 mg intravenously once daily for 5 consecutive days in participants with relapse.
  Interventions: Dietary Supplement: D-aspartate; Biological: IFN beta-1a; Drug: Methylprednisolone
- Placebo + IFN beta-1a + Methylprednisolone (Placebo Comparator): Participants received placebo matched to D-aspartate once daily in the form of oral solution for 24 weeks along with IFN beta-1a subcutaneously (sc) at a dose of 44 microgram (mcg) three times a week (TIW) in participants without relapse and IFN beta-1a sc TIW plus Methylprednisolone 1000 mg intravenously once daily for 5 consecutive days in participants with relapse.
  Interventions: Drug: Placebo; Biological: IFN beta-1a; Drug: Methylprednisolone

INTERVENTIONS:
Dietary Supplement: D-aspartate — D-aspartate 2660 milligram (mg) once daily in the form of oral solution for 24 weeks.
  Arms: D-aspartate + IFN beta-1a + Methylprednisolone
Drug: Placebo — Placebo matched to D-aspartate once daily in the form of oral solution for 24 weeks.
  Arms: Placebo + IFN beta-1a + Methylprednisolone
Biological: IFN beta-1a — IFN beta-1a was administered subcutaneously at a dose of 44 microgram (mcg) three times a week for 24 weeks.
Drug: Methylprednisolone — Methylprednisolone 1000 mg was administered intravenously once daily for 5 consecutive days.

SUMMARY:
The purpose of this study was to evaluate the improvement in spontaneous recovery from clinical deficits at the time of an acute relapse in RR-MS participants already receiving interferon (IFN) beta 1a with D-aspartate (versus placebo) as add-on therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participants with RR-MS, according to the revised McDonald Criteria (2010)
* Participants with an expanded disability status scale (EDSS) score between 0 and 3 before screening visit and before relapse
* Participants receiving treatment with IFN beta 1a 44 mcg three times a week for at least 6 months but for no more than 10 years before the screening visit
* Female participants must be neither pregnant nor breastfeeding and must lack childbearing potential
* Participants willing and able to comply with the protocol for the total duration of the study
* Participants able to understand the purposes and the risks of the study
* Participants have signed the appropriate written informed consent form, approved by the Independent Ethics Committee (IEC), prior to the performance of any study activities
* For MS participants with relapse:
* Deterioration of at least one step in a relevant Functional Systems Scale (FSS) or an increase in EDSS of 1 point or more compatible, according to physician's judgment, with the therapy prosecution
* Relapse started within maximum 5 days before the inclusion in the study
* MS participants without relapse with clinically stable RR-MS

Exclusion Criteria:

* Participants with diagnosis of primary progressive MS (PP-MS)
* Participants have any disease other than MS that could better explain his/her signs and symptoms
* Participants with any comorbidity with diseases that might alter synaptic plasticity (example Parkinson Disease, Alzheimer Disease, Stroke)
* Participants receiving concomitant treatment with drugs that may alter synaptic plasticity (example, cannabinoids)
* Participants with history or presence of any unstable medical condition (tumor or chronic infection or severe life threatening infection within the last 6 months)
* Participants who have received any corticosteroids therapy within 3 months prior to the screening
* Participants with any concomitant disease that may require chronic treatment with systemic corticosteroids or immunosuppressive agents during the course of the study
* Participants who have received any immunosuppressive agents other to corticosteroids, as monotherapy or combination therapy within 3 months prior to the screening visit
* Participants with history or currently active primary or secondary immunodeficiency
* Participants with inadequate liver function, defined by alanine aminotransferase (ALT) > 3 * upper limit of normal (ULN), or alkaline phosphatase (AP) > 2 * ULN, or total bilirubin > 2 * ULN if associated with any elevation of ALT or AP
* Participants with inadequate bone marrow reserve, defined as a white blood cell count less than 0.5 * lower limit of normal (LLN)
* Participants with moderate to severe renal impairment
* Participants unable to complete an magnetic resonance imaging (MRI) (contraindications for MRI include but are not restricted to weight >=140 kilogram (kg), pacemaker, cochlear implants, presence of foreign substances in the eye, intracranial vascular clips, surgery within 6 weeks of entry into the study, coronary stent implanted within 8 weeks prior to the time of the intended MRI, etc)
* Participants with contraindication to gadolinium (Gd) can be enrolled into the study but cannot receive Gd contrast dyes during their MRI scans
* Participants receiving supplements that, in the Investigator's opinion, may affect the evaluation of fatigue
* Participants with any known contraindications or hypersensitivity to D-aspartate or any excipient
* Participants with any other significant disease that in the Investigator's opinion would impede study assessments or endanger the participant
* Female participants with positive pregnancy test at baseline or participants with active project of pregnancy during the study
* Participants with legal incapacity or limited legal capacity
* Participants have participated in any other investigational study within 8 weeks before the screening visit

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-01-11 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (17):
- Italy (17):
  - Ospedale Binaghi, Università di Cagliari,ASL 8, Cagliari
  - Ospedale Clinicizzato SS. Annunziata, Chieti
  - Azienda Socio Sanitaria Territoriale della Valle Olona (presidio di Gallarate), Gallarate
  - Azienda Ospedaliero Universitaria San Martino, Genova
  - Ospedale P.A.Micone, Genova
  - Ospedale San Raffaele, Milan
  - A.O.U. Federico II, Napoli
  - Azienda Ospedaliera di Rilievo Nazionale A. CardarelliAzienda Ospedaliera di Rilievo Nazionale A. Cardarelli, Napoli
  - Seconda Università degli Studi di Napoli, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - I.R.C.C.S. Neuromed-Istituto Neurologico Mediterraneo, Pozzilli
  - Azienda Ospedaliera San Camillo Forlanini, Roma
  - Azienda Ospedaliera Sant'Andrea-Università di Roma La Sapienza, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome
  - Ospedale S. Paolo, Savona
  - Azienda Ospedaliero Universitaria Ospedali Riuniti, Torrette Di Ancona

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Started | 5 | 2
Completed | 4 | 1
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone | Total
Number analyzed (Participants) | 5 | 2 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 5 | 2 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Change From Baseline in Multiple Sclerosis Related Disability Measured by Expanded Disability Status Scale (EDSS) at Week 8
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with Multiple Sclerosis (MS). It assesses the 8 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder, cerebral and other) as well as ambulation. EDSS overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: Baseline, Week 8
Population: Full analysis set included all participants enrolled into the study and assigned to the randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
Participants | 1 | 0

2. Secondary Outcome: Number of Participants With Change From Baseline in Multiple Sclerosis Related Disability Measured by Expanded Disability Status Scale (EDSS) at Week 12 and 24
Description: EDSS is an ordinal scale in half-point increments that qualifies disability in participants with Multiple Sclerosis. It assesses the 8 functional systems (visual, brainstem, pyramidal, cerebellar, sensory, bowel/bladder, cerebral and other) as well as ambulation. EDSS overall score ranging from 0 (normal) to 10 (death due to MS).
Time Frame: Baseline, Week 12 and 24
Population: Full analysis set included all participants enrolled into the study and assigned to the randomized treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
Participants
  Week 12 | 1 | 0
  Week 24 | 1 | 0

3. Secondary Outcome: 25-foot Timed Walk (25-FWT) to Measure Multiple Sclerosis Related Disability and Cognitive Impairment
Description: The Timed 25-Foot Walk is a quantitative measure of lower extremity function. The participants is directed to one end of a clearly marked 25-foot (7.62 m) course and is instructed to walk 25 feet (7.62 meter) as quickly as possible, but safely. The task is immediately administered again by having the participant walk back the same distance. Participants may use assistive devices when doing this task. The test scores were the time in seconds it took to walk the 25 feet. The data for the 25-FWT is reported for the 2 completed trials. Participant wise data was reported for this outcome.
Time Frame: At Week 8, 12 and 24
Population: Full analysis set included all participants enrolled into the study and assigned to the randomized treatment. No summary analysis was done as study was prematurely terminated due to slow recruitment rate and participant wise data are reported. Here, "number analyzed" signifies specific participant evaluated in respective arm at specified timepoint.
Measure: Number; unit: Seconds
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
Seconds
  Participant 1: Trial 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 8 | 13.1 |
  Participant 1: Trial 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 8 | 12.4 |
  Participant 2: Trial 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 2: Trial 1: Week 8 | 12.7 |
  Participant 2: Trial 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 2: Trial 2: Week 8 | 12.6 |
  Participant 3: Trial 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 8 | 17.4 |
  Participant 3: Trial 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 8 | 16.3 |
  Participant 4: Trial 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 8 | 11.3 |
  Participant 4: Trial 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 8 | 10.9 |
  Participant 5: Trial 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 8 | 5.6 |
  Participant 5: Trial 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 8 | 5.7 |
  Participant 6: Trial 1: Week 8: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 1: Week 8 |  | 16.1
  Participant 6: Trial 2: Week 8: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 2: Week 8 |  | 14.3
  Participant 7: Trial 1: Week 8: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 8 |  | 9.3
  Participant 7: Trial 2: Week 8: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 8 |  | 8.9
  Participant 1: Trial 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 12 | 13.1 |
  Participant 1: Trial 2: Week 12: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 12 | 13.8 |
  Participant 3: Trial 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 12 | 17.1 |
  Participant 3: Trial 2: Week 12: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 12 | 15.8 |
  Participant 4: Trial 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 12 | 10.9 |
  Participant 4: Trial 2: Week 12: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 12 | 10.2 |
  Participant 5: Trial 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 12 | 5.7 |
  Participant 5: Trial 2: Week 12: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 12 | 5.6 |
  Participant 6: Trial 1: Week 12: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 1: Week 12 |  | 12.7
  Participant 6: Trial 2: Week 12: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 2: Week 12 |  | 12.3
  Participant 7: Trial 1: Week 12: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 12 |  | 12.4
  Participant 7: Trial 2: Week 12: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 12 |  | 11.8
  Participant 1: Trial 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 24 | 11.8 |
  Participant 1: Trial 2: Week 24: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 24 | 11.5 |
  Participant 3: Trial 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 24 | 8.6 |
  Participant 3: Trial 2: Week 24: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 24 | 9.3 |
  Participant 4: Trial 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 24 | 11.4 |
  Participant 4: Trial 2: Week 24: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 24 | 11.5 |
  Participant 5: Trial 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 24 | 5.0 |
  Participant 5: Trial 2: Week 24: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 24 | 5.3 |
  Participant 7: Trial 1: Week 24: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 24 |  | 10.1
  Participant 7: Trial 2: Week 24: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 24 |  | 9.8

4. Secondary Outcome: 9 Hole Peg Test (9HPT) to Measure Multiple Sclerosis Related Disability and Cognitive Impairment
Description: The 9HPT is a brief, standardized, quantitative test of upper extremity function. The participant picks up 9 pegs puts them in a block containing nine empty holes, and, once they are in the holes, removes them again as quickly as possible one at a time. The total time to complete the task is recorded. Two consecutive trials with the dominant hand are immediately followed by two consecutive trials with the non-dominant hand. The data for the 29HPT is reported for the 2 completed trials. Participant wise data was reported for this outcome.
Time Frame: Week 8, 12 and 24
Population: as for outcome 3
Measure: Number; unit: Seconds
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
Seconds
  Participant 1: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 8: Dominant hand | 22.1 |
  Participant 1: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 8: Dominant hand | 21.1 |
  Participant 2: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 2: Trial 1: Week 8: Dominant hand | 18.7 |
  Participant 2: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 2: Trial 2: Week 8: Dominant hand | 17.6 |
  Participant 3: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 8: Dominant hand | 19.7 |
  Participant 3: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 8: Dominant hand | 16.3 |
  Participant 4: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 8: Dominant hand | 17.8 |
  Participant 4: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 8: Dominant hand | 17.2 |
  Participant 5: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 8: Dominant hand | 22.6 |
  Participant 5: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 8: Dominant hand | 25.5 |
  Participant 6: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 1: Week 8: Dominant hand |  | 17.5
  Participant 6: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 2: Week 8: Dominant hand |  | 17.2
  Participant 7: Trial 1: Week 8: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 8: Dominant hand |  | 31.9
  Participant 7: Trial 2: Week 8: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 8: Dominant hand |  | 9.5
  Participant 1: Trial 1: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 12: Dominant hand | 24.2 |
  Participant 1: Trial 2: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 12: Dominant hand | 22.0 |
  Participant 3: Trial 1: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 12: Dominant hand | 17.6 |
  Participant 3: Trial 2: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 12: Dominant hand | 17.8 |
  Participant 4: Trial 1: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 12: Dominant hand | 16.8 |
  Participant 4: Trial 2: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 12: Dominant hand | 16.1 |
  Participant 5: Trial 1: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 12: Dominant hand | 25.3 |
  Participant 5: Trial 2: Week 12: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 12: Dominant hand | 23.2 |
  Participant 6: Trial 1: Week 12: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 1: Week 12: Dominant hand |  | 21.1
  Participant 6: Trial 2: Week 12: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 2: Week 12: Dominant hand |  | 17.9
  Participant 7: Trial 1: Week 12: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 12: Dominant hand |  | 31.6
  Participant 7: Trial 2: Week 12: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 12: Dominant hand |  | 29.8
  Participant 1: Trial 1: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 24: Dominant hand | 22.0 |
  Participant 1: Trial 2: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 24: Dominant hand | 21.5 |
  Participant 3: Trial 1: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 24: Dominant hand | 18.8 |
  Participant 3: Trial 2: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 24: Dominant hand | 18.1 |
  Participant 4: Trial 1: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 24: Dominant hand | 17.2 |
  Participant 4: Trial 2: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 24: Dominant hand | 16.7 |
  Participant 5: Trial 1: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 24: Dominant hand | 27.4 |
  Participant 5: Trial 2: Week 24: Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 24: Dominant hand | 24.6 |
  Participant 7: Trial 1: Week 24: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 24: Dominant hand |  | 32.6
  Participant 7: Trial 2: Week 24: Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 24: Dominant hand |  | 30.8
  Participant 1: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 8: Non-Dominant hand | 25.2 |
  Participant 1: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 8: Non-Dominant hand | 25.3 |
  Participant 2: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 2: Trial 1: Week 8: Non-Dominant hand | 18.9 |
  Participant 2: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 2: Trial 2: Week 8: Non-Dominant hand | 17.3 |
  Participant 3: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 8: Non-Dominant hand | 21.4 |
  Participant 3: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 8: Non-Dominant hand | 20.7 |
  Participant 4: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 8: Non-Dominant hand | 18.9 |
  Participant 4: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 8: Non-Dominant hand | 19.7 |
  Participant 5: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 8: Non-Dominant hand | 22.0 |
  Participant 5: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 8: Non-Dominant hand | 20.8 |
  Participant 6: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 1: Week 8: Non-Dominant hand |  | 19.5
  Participant 6: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 2: Week 8: Non-Dominant hand |  | 19.9
  Participant 7: Trial 1: Week 8: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 8: Non-Dominant hand |  | 22.0
  Participant 7: Trial 2: Week 8: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 8: Non-Dominant hand |  | 21.1
  Participant 1: Trial 1: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 12: Non-Dominant hand | 22.8 |
  Participant 1: Trial 2: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 12: Non-Dominant hand | 19.8 |
  Participant 3: Trial 1: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 12: Non-Dominant hand | 20.8 |
  Participant 3: Trial 2: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 12: Non-Dominant hand | 22.5 |
  Participant 4: Trial 1: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 12: Non-Dominant hand | 17.3 |
  Participant 4: Trial 2: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 12: Non-Dominant hand | 17.5 |
  Participant 5: Trial 1: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 12: Non-Dominant hand | 22.8 |
  Participant 5: Trial 2: Week 12: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 12: Non-Dominant hand | 23.7 |
  Participant 6: Trial 1: Week 12: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 1: Week 12: Non-Dominant hand |  | 20.6
  Participant 6: Trial 2: Week 12: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 6: Trial 2: Week 12: Non-Dominant hand |  | 20.4
  Participant 7: Trial 1: Week 12: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 12: Non-Dominant hand |  | 24.5
  Participant 7: Trial 2: Week 12: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 12: Non-Dominant hand |  | 25.7
  Participant 1: Trial 1: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 1: Week 24: Non-Dominant hand | 22.4 |
  Participant 1: Trial 2: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 1: Trial 2: Week 24: Non-Dominant hand | 20.5 |
  Participant 3: Trial 1: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 1: Week 24: Non-Dominant hand | 20.1 |
  Participant 3: Trial 2: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 3: Trial 2: Week 24: Non-Dominant hand | 18.4 |
  Participant 4: Trial 1: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 1: Week 24: Non-Dominant hand | 18.1 |
  Participant 4: Trial 2: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 4: Trial 2: Week 24: Non-Dominant hand | 18.3 |
  Participant 5: Trial 1: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 1: Week 24: Non-Dominant hand | 25.8 |
  Participant 5: Trial 2: Week 24: Non-Dominant hand: number analyzed (Participants) | 1 | 0
  Participant 5: Trial 2: Week 24: Non-Dominant hand | 22.7 |
  Participant 7: Trial 1: Week 24: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 1: Week 24: Non-Dominant hand |  | 24.1
  Participant 7: Trial 2: Week 24: Non-Dominant hand: number analyzed (Participants) | 0 | 1
  Participant 7: Trial 2: Week 24: Non-Dominant hand |  | 23.6

5. Secondary Outcome: Symbol Digit Modalities Test to Measure Multiple Sclerosis Related Disability and Cognitive Impairment
Description: Symbol digit modalities test is to evaluate neurocognitive functions. This measure involves a coding key consisting of 9 abstract symbols, each paired with a number ranging from 1 to 9. The participants is required to scan the key and write down the number corresponding to each symbol as fast as possible. The number of correct substitution within 90 seconds is recorded. In the written version of the test the participants fills in the numbers that correspond to the symbols. The score is the number of correctly coded items from 0-110 in 90 seconds. A higher score indicates better performance. Participant wise data was reported for this outcome.
Time Frame: At Week 8, 12 and 24
Population: as for outcome 3
Measure: Number; unit: units on a scale
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
units on a scale
  Participant 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 1: Week 8 | 38 |
  Participant 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 2: Week 8 | 43 |
  Participant 3: Week 8: number analyzed (Participants) | 1 | 0
  Participant 3: Week 8 | 48 |
  Participant 4: Week 8: number analyzed (Participants) | 1 | 0
  Participant 4: Week 8 | 66 |
  Participant 5: Week 8: number analyzed (Participants) | 1 | 0
  Participant 5: Week 8 | 46 |
  Participant 6: Week 8: number analyzed (Participants) | 0 | 1
  Participant 6: Week 8 |  | 56
  Participant 7: Week 8: number analyzed (Participants) | 0 | 1
  Participant 7: Week 8 |  | 43
  Participant 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 1: Week 12 | 48 |
  Participant 3: Week 12: number analyzed (Participants) | 1 | 0
  Participant 3: Week 12 | 44 |
  Participant 4: Week 12: number analyzed (Participants) | 1 | 0
  Participant 4: Week 12 | 68 |
  Participant 5: Week 12: number analyzed (Participants) | 1 | 0
  Participant 5: Week 12 | 44 |
  Participant 6: Week 12: number analyzed (Participants) | 0 | 1
  Participant 6: Week 12 |  | 46
  Participant 7: Week 12: number analyzed (Participants) | 0 | 1
  Participant 7: Week 12 |  | 43
  Participant 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 1: Week 24 | 50 |
  Participant 3: Week 24: number analyzed (Participants) | 1 | 0
  Participant 3: Week 24 | 51 |
  Participant 4: Week 24: number analyzed (Participants) | 1 | 0
  Participant 4: Week 24 | 70 |
  Participant 5: Week 24: number analyzed (Participants) | 1 | 0
  Participant 5: Week 24 | 39 |
  Participant 7: Week 24: number analyzed (Participants) | 0 | 1
  Participant 7: Week 24 |  | 55

6. Secondary Outcome: Low Contrast Letter Visual Acuity Test to Measure Multiple Sclerosis Related Disability and Cognitive Impairment
Description: Visual acuity is measured under low contrast conditions (10% contrast relative to the chart background) at object testing distances of 10 feets and is reported as the number of letters read correctly (ranging from 0 to 10 letters). The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly indicates that vision has improved. Participant wise data was reported for this outcome.
Time Frame: Week 8, 12 and 24
Population: Full analysis set. No summary analysis was done as study was prematurely terminated due to slow recruitment rate and participant wise data are reported. Here, "Number of participants analyzed" signifies those who were evaluable for this endpoint and "number analyzed" signifies specific participant evaluated in respective arm at specified timepoint.
Measure: Number; unit: Letters read correctly
Units Other Than Participants: eye
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 4 | 2
Number analyzed (eye) | 8 | 4
Letters read correctly
  Participant 1: Week 8: Left eye: number analyzed (Participants) | 1 | 0
  Participant 1: Week 8: Left eye: number analyzed (eye) | 1 | 0
  Participant 1: Week 8: Left eye | 4 |
  Participant 2: Week 8: Left eye: number analyzed (Participants) | 1 | 0
  Participant 2: Week 8: Left eye: number analyzed (eye) | 1 | 0
  Participant 2: Week 8: Left eye | 8 |
  Participant 3: Week 8: Left eye: number analyzed (Participants) | 1 | 0
  Participant 3: Week 8: Left eye: number analyzed (eye) | 1 | 0
  Participant 3: Week 8: Left eye | 8 |
  Participant 4: Week 8: Left eye: number analyzed (Participants) | 1 | 0
  Participant 4: Week 8: Left eye: number analyzed (eye) | 1 | 0
  Participant 4: Week 8: Left eye | 8 |
  Participant 6: Week 8: Left eye: number analyzed (Participants) | 0 | 1
  Participant 6: Week 8: Left eye: number analyzed (eye) | 0 | 1
  Participant 6: Week 8: Left eye |  | 8
  Participant 7: Week 8: Left eye: number analyzed (Participants) | 0 | 1
  Participant 7: Week 8: Left eye: number analyzed (eye) | 0 | 1
  Participant 7: Week 8: Left eye |  | 8
  Participant 1: Week 12: Left eye: number analyzed (Participants) | 1 | 0
  Participant 1: Week 12: Left eye: number analyzed (eye) | 1 | 0
  Participant 1: Week 12: Left eye | 2 |
  Participant 3: Week 12: Left eye: number analyzed (Participants) | 1 | 0
  Participant 3: Week 12: Left eye: number analyzed (eye) | 1 | 0
  Participant 3: Week 12: Left eye | 10 |
  Participant 4: Week 12: Left eye: number analyzed (Participants) | 1 | 0
  Participant 4: Week 12: Left eye: number analyzed (eye) | 1 | 0
  Participant 4: Week 12: Left eye | 8 |
  Participant 6: Week 12: Left eye: number analyzed (Participants) | 0 | 1
  Participant 6: Week 12: Left eye: number analyzed (eye) | 0 | 1
  Participant 6: Week 12: Left eye |  | 8
  Participant 7: Week 12: Left eye: number analyzed (Participants) | 0 | 1
  Participant 7: Week 12: Left eye: number analyzed (eye) | 0 | 1
  Participant 7: Week 12: Left eye |  | 9
  Participant 1: Week 24: Left eye: number analyzed (Participants) | 1 | 0
  Participant 1: Week 24: Left eye: number analyzed (eye) | 1 | 0
  Participant 1: Week 24: Left eye | 3 |
  Participant 3: Week 24: Left eye: number analyzed (Participants) | 1 | 0
  Participant 3: Week 24: Left eye: number analyzed (eye) | 1 | 0
  Participant 3: Week 24: Left eye | 10 |
  Participant 4: Week 24: Left eye: number analyzed (Participants) | 1 | 0
  Participant 4: Week 24: Left eye: number analyzed (eye) | 1 | 0
  Participant 4: Week 24: Left eye | 10 |
  Participant 7: Week 24: Left eye: number analyzed (Participants) | 0 | 1
  Participant 7: Week 24: Left eye: number analyzed (eye) | 0 | 1
  Participant 7: Week 24: Left eye |  | 8
  Participant 1: Week 8: Right eye: number analyzed (Participants) | 1 | 0
  Participant 1: Week 8: Right eye: number analyzed (eye) | 1 | 0
  Participant 1: Week 8: Right eye | 4 |
  Participant 2: Week 8: Right eye: number analyzed (Participants) | 1 | 0
  Participant 2: Week 8: Right eye: number analyzed (eye) | 1 | 0
  Participant 2: Week 8: Right eye | 8 |
  Participant 3: Week 8: Right eye: number analyzed (Participants) | 1 | 0
  Participant 3: Week 8: Right eye: number analyzed (eye) | 1 | 0
  Participant 3: Week 8: Right eye | 2 |
  Participant 4: Week 8: Right eye: number analyzed (Participants) | 1 | 0
  Participant 4: Week 8: Right eye: number analyzed (eye) | 1 | 0
  Participant 4: Week 8: Right eye | 7 |
  Participant 6: Week 8: Right eye: number analyzed (Participants) | 0 | 1
  Participant 6: Week 8: Right eye: number analyzed (eye) | 0 | 1
  Participant 6: Week 8: Right eye |  | 8
  Participant 7: Week 8: Right eye: number analyzed (Participants) | 0 | 1
  Participant 7: Week 8: Right eye: number analyzed (eye) | 0 | 1
  Participant 7: Week 8: Right eye |  | 8
  Participant 1: Week 12: Right eye: number analyzed (Participants) | 1 | 0
  Participant 1: Week 12: Right eye: number analyzed (eye) | 1 | 0
  Participant 1: Week 12: Right eye | 8 |
  Participant 3: Week 12: Right eye: number analyzed (Participants) | 1 | 0
  Participant 3: Week 12: Right eye: number analyzed (eye) | 1 | 0
  Participant 3: Week 12: Right eye | 10 |
  Participant 4: Week 12: Right eye: number analyzed (Participants) | 1 | 0
  Participant 4: Week 12: Right eye: number analyzed (eye) | 1 | 0
  Participant 4: Week 12: Right eye | 7 |
  Participant 6: Week 12: Right eye: number analyzed (Participants) | 0 | 1
  Participant 6: Week 12: Right eye: number analyzed (eye) | 0 | 1
  Participant 6: Week 12: Right eye |  | 8
  Participant 7: Week 12: Right eye: number analyzed (Participants) | 0 | 1
  Participant 7: Week 12: Right eye: number analyzed (eye) | 0 | 1
  Participant 7: Week 12: Right eye |  | 9
  Participant 1: Week 24: Right eye: number analyzed (Participants) | 1 | 0
  Participant 1: Week 24: Right eye: number analyzed (eye) | 1 | 0
  Participant 1: Week 24: Right eye | 8 |
  Participant 3: Week 24: Right eye: number analyzed (Participants) | 1 | 0
  Participant 3: Week 24: Right eye: number analyzed (eye) | 1 | 0
  Participant 3: Week 24: Right eye | 10 |
  Participant 4: Week 24: Right eye: number analyzed (Participants) | 1 | 0
  Participant 4: Week 24: Right eye: number analyzed (eye) | 1 | 0
  Participant 4: Week 24: Right eye | 10 |
  Participant 7: Week 24: Right eye: number analyzed (Participants) | 0 | 1
  Participant 7: Week 24: Right eye: number analyzed (eye) | 0 | 1
  Participant 7: Week 24: Right eye |  | 8

7. Secondary Outcome: Modified Fatigue Impact Scale (MFIS) Score to Measure Fatigue at Week 8, 12 and 24
Description: MFIS is a structured, self-report questionnaire consisting of 21 items assessing the effects of fatigue. All 21 items are scaled 0 to 4, with higher scores indicating a greater impact of fatigue on participant's activities. The Total MFIS score ranges from 0 to 84. A score of 0 indicates fatigue has no impact on activities and the high-end score indicates fatigue has extreme impact on activities. Participant wise data was reported for this outcome.
Time Frame: Week 8, 12 and 24
Population: as for outcome 3
Measure: Number; unit: units on a scale
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
units on a scale
  Participant 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 1: Week 8 | 8 |
  Participant 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 2: Week 8 | 27 |
  Participant 3: Week 8: number analyzed (Participants) | 1 | 0
  Participant 3: Week 8 | 15 |
  Participant 4: Week 8: number analyzed (Participants) | 1 | 0
  Participant 4: Week 8 | 2 |
  Participant 5: Week 8: number analyzed (Participants) | 1 | 0
  Participant 5: Week 8 | 18 |
  Participant 6: Week 8: number analyzed (Participants) | 0 | 1
  Participant 6: Week 8 |  | 27
  Participant 7: Week 8: number analyzed (Participants) | 0 | 1
  Participant 7: Week 8 |  | 29
  Participant 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 1: Week 12 | 6 |
  Participant 3: Week 12: number analyzed (Participants) | 1 | 0
  Participant 3: Week 12 | 12 |
  Participant 4: Week 12: number analyzed (Participants) | 1 | 0
  Participant 4: Week 12 | 12 |
  Participant 5: Week 12: number analyzed (Participants) | 1 | 0
  Participant 5: Week 12 | 15 |
  Participant 6: Week 12: number analyzed (Participants) | 0 | 1
  Participant 6: Week 12 |  | 27
  Participant 7: Week 12: number analyzed (Participants) | 0 | 1
  Participant 7: Week 12 |  | 30
  Participant 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 1: Week 24 | 10 |
  Participant 3: Week 24: number analyzed (Participants) | 1 | 0
  Participant 3: Week 24 | 48 |
  Participant 4: Week 24: number analyzed (Participants) | 1 | 0
  Participant 4: Week 24 | 12 |
  Participant 5: Week 24: number analyzed (Participants) | 1 | 0
  Participant 5: Week 24 | 15 |
  Participant 7: Week 24: number analyzed (Participants) | 0 | 1
  Participant 7: Week 24 |  | 43

8. Secondary Outcome: Fatigue Severity Scale (FSS) Score to Measure Fatigue by at Week 8, 12 and 24
Description: Fatigue Severity Scale (FSS) is a method of evaluating fatigue in multiple sclerosis and is designed to differentiate fatigue from clinical depression, since both share some of the same symptoms. The Fatigue Severity Scale is a 9-item questionnaire developed to assess the level of fatigue due to neurological disease, were each assessed on a 1-7 scale (1= no fatigue and 7= severe fatigue). The total score was calculated as the average of individual 9-items and ranged from 1 to 7 with a higher value indicating greater impairment due to fatigue. Participant wise data was reported for this outcome.
Time Frame: Week 8, 12 and 24
Population: as for outcome 3
Measure: Number; unit: units on a scale
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 5 | 2
units on a scale
  Participant 1: Week 8: number analyzed (Participants) | 1 | 0
  Participant 1: Week 8 | 1.2 |
  Participant 2: Week 8: number analyzed (Participants) | 1 | 0
  Participant 2: Week 8 | 2.6 |
  Participant 3: Week 8: number analyzed (Participants) | 1 | 0
  Participant 3: Week 8 | 1.7 |
  Participant 4: Week 8: number analyzed (Participants) | 1 | 0
  Participant 4: Week 8 | 1.1 |
  Participant 5: Week 8: number analyzed (Participants) | 1 | 0
  Participant 5: Week 8 | 1 |
  Participant 6: Week 8: number analyzed (Participants) | 0 | 1
  Participant 6: Week 8 |  | 4.3
  Participant 7: Week 8: number analyzed (Participants) | 0 | 1
  Participant 7: Week 8 |  | 2.2
  Participant 1: Week 12: number analyzed (Participants) | 1 | 0
  Participant 1: Week 12 | 1.3 |
  Participant 3: Week 12: number analyzed (Participants) | 1 | 0
  Participant 3: Week 12 | 2.6 |
  Participant 4: Week 12: number analyzed (Participants) | 1 | 0
  Participant 4: Week 12 | 2 |
  Participant 5: Week 12: number analyzed (Participants) | 1 | 0
  Participant 5: Week 12 | 1 |
  Participant 6: Week 12: number analyzed (Participants) | 0 | 1
  Participant 6: Week 12 |  | 4.1
  Participant 7: Week 12: number analyzed (Participants) | 0 | 1
  Participant 7: Week 12 |  | 4.1
  Participant 1: Week 24: number analyzed (Participants) | 1 | 0
  Participant 1: Week 24 | 1.3 |
  Participant 3: Week 24: number analyzed (Participants) | 1 | 0
  Participant 3: Week 24 | 2.8 |
  Participant 4: Week 24: number analyzed (Participants) | 1 | 0
  Participant 4: Week 24 | 2 |
  Participant 5: Week 24: number analyzed (Participants) | 1 | 0
  Participant 5: Week 24 | 1.1 |
  Participant 7: Week 24: number analyzed (Participants) | 0 | 1
  Participant 7: Week 24 |  | 3.3

9. Secondary Outcome: Long Term Potentiation Measured by Transcranial Magnetic Stimulation (TMS)
Description: TMS is an electrophysiological technique that was used to measure neurologic changes associated with recovery from stroke via alterations in the excitability of the motor system. Motor threshold measures reflect global excitability of the corticospinal pathway, including large pyramidal cells, excitatory/inhibitory interneurons, and spinal motor neurons. Long term potentiation can be measured non invasively and painlessly, in awake humans through transcranial magnetic stimulation (TMS). TMS uses high intensity, brief duration, magnetic fields that, when applied on the scalp, can activate neurons within a small focal region of the cerebral cortex, through electromagnetic induction. Motor Evoked Potentials (MEP) amplitudes elicited by single TMS pulses of increasing intensity (110, 120 and 130% of the Resting Motor Threshold [RMT]) will be measured to calculate recruitment curves of the motor cortex. Participant wise data was reported for this outcome.
Time Frame: Baseline (0 minute) and Post-Baseline (15 minutes) at Week 8
Population: Full analysis set. No summary analysis was done as study was prematurely terminated due to slow recruitment rate and participant wise data are reported. Here, "Number of participants analyzed" signifies those who were evaluated for this endpoint and "number analyzed" signifies specific participant evaluated in respective arm.
Measure: Number; unit: millivolts
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 2 | 2
millivolts
  Participants 1: Week 8 (Baseline): 110% RMT: number analyzed (Participants) | 1 | 0
  Participants 1: Week 8 (Baseline): 110% RMT | 30 |
  Participants 1: Week 8 (Baseline): 120% RMT: number analyzed (Participants) | 1 | 0
  Participants 1: Week 8 (Baseline): 120% RMT | 105 |
  Participants 1: Week 8 (Baseline): 130% RMT: number analyzed (Participants) | 1 | 0
  Participants 1: Week 8 (Baseline): 130% RMT | 142 |
  Participants 1: Week 8 (Post-baseline): 110% RMT: number analyzed (Participants) | 1 | 0
  Participants 1: Week 8 (Post-baseline): 110% RMT | 39 |
  Participants 1: Week 8 (Post-baseline): 120% RMT: number analyzed (Participants) | 1 | 0
  Participants 1: Week 8 (Post-baseline): 120% RMT | 128 |
  Participants 1: Week 8 (Post-baseline): 130% RMT: number analyzed (Participants) | 1 | 0
  Participants 1: Week 8 (Post-baseline): 130% RMT | 154 |
  Participants 3: Week 8 (Baseline): 110% RMT: number analyzed (Participants) | 1 | 0
  Participants 3: Week 8 (Baseline): 110% RMT | 23 |
  Participants 3: Week 8 (Baseline): 120% RMT: number analyzed (Participants) | 1 | 0
  Participants 3: Week 8 (Baseline): 120% RMT | 95 |
  Participants 3: Week 8 (Baseline): 130% RMT: number analyzed (Participants) | 1 | 0
  Participants 3: Week 8 (Baseline): 130% RMT | 115 |
  Participants 3: Week 8 (Post-baseline): 110% RMT: number analyzed (Participants) | 1 | 0
  Participants 3: Week 8 (Post-baseline): 110% RMT | 31 |
  Participants 3: Week 8 (Post-baseline): 120% RMT: number analyzed (Participants) | 1 | 0
  Participants 3: Week 8 (Post-baseline): 120% RMT | 103 |
  Participants 3: Week 8 (Post-baseline): 130% RMT: number analyzed (Participants) | 1 | 0
  Participants 3: Week 8 (Post-baseline): 130% RMT | 118 |
  Participants 6: Week 8 (Baseline): 110% RMT: number analyzed (Participants) | 0 | 1
  Participants 6: Week 8 (Baseline): 110% RMT |  | 28
  Participants 6: Week 8 (Baseline): 120% RMT: number analyzed (Participants) | 0 | 1
  Participants 6: Week 8 (Baseline): 120% RMT |  | 83
  Participants 6: Week 8 (Baseline): 130% RMT: number analyzed (Participants) | 0 | 1
  Participants 6: Week 8 (Baseline): 130% RMT |  | 118
  Participants 6: Week 8 (Post-baseline): 110% RMT: number analyzed (Participants) | 0 | 1
  Participants 6: Week 8 (Post-baseline): 110% RMT |  | 26
  Participants 6: Week 8 (Post-baseline): 120% RMT: number analyzed (Participants) | 0 | 1
  Participants 6: Week 8 (Post-baseline): 120% RMT |  | 91
  Participants 6: Week 8 (Post-baseline): 130% RMT: number analyzed (Participants) | 0 | 1
  Participants 6: Week 8 (Post-baseline): 130% RMT |  | 125
  Participants 7: Week 8 (Baseline): 110% RMT: number analyzed (Participants) | 0 | 1
  Participants 7: Week 8 (Baseline): 110% RMT |  | 33
  Participants 7: Week 8 (Baseline): 120% RMT: number analyzed (Participants) | 0 | 1
  Participants 7: Week 8 (Baseline): 120% RMT |  | 140
  Participants 7: Week 8 (Baseline): 130% RMT: number analyzed (Participants) | 0 | 1
  Participants 7: Week 8 (Baseline): 130% RMT |  | 149
  Participants 7: Week 8 (Post-baseline): 110% RMT: number analyzed (Participants) | 0 | 1
  Participants 7: Week 8 (Post-baseline): 110% RMT |  | 30
  Participants 7: Week 8 (Post-baseline): 120% RMT: number analyzed (Participants) | 0 | 1
  Participants 7: Week 8 (Post-baseline): 120% RMT |  | 135
  Participants 7: Week 8 (Post-baseline): 130% RMT: number analyzed (Participants) | 0 | 1
  Participants 7: Week 8 (Post-baseline): 130% RMT |  | 138

10. Secondary Outcome: Number of Treated Participants With Immune-metabolic Response of Lymphocytes
Description: Treated participants with immune-metabolic response (glycolysis, mitochondrial respiration, fatty acids oxidation and circulating adipocytokines) of lymphocytes were to be reported.
Time Frame: Baseline, Week 8 and 12
Population: Data was not collected since the study was prematurely terminated, due to slow recruitment rate.
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to 292 days; Participants were assessed for adverse events for the entire study
Arm/Group | D-aspartate + IFN Beta-1a + Methylprednisolone | Placebo + IFN Beta-1a + Methylprednisolone
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 3/5 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | D-aspartate + IFN Beta-1a + Methylprednisolone (N=5) | Placebo + IFN Beta-1a + Methylprednisolone (N=2)
Hypersexuality (Reproductive system and breast disorders) | 1 | 0
Flu-like symptoms (Infections and infestations) | 1 | 1
Weight gain (General disorders) | 1 | 0
Pain in the left thigh (General disorders) | 1 | 0
Periorbital pain (Eye disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study was prematurely terminated, due to slow recruitment rate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT03387046/Prot_SAP_000.pdf